CLINICAL TRIAL: NCT01977365
Title: Effectiveness of Child Centered Counseling on Child Nutrition Status. A Cluster Randomized Trial in Rural Burkina Faso.
Brief Title: Effectiveness of Child Centered Counseling on Child Nutrition Status
Acronym: LUCOMAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Laetitia Ouedraogo, Chargée de Recherche, Institut de Recherche en Sciences de la Sante, Burkina Faso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRSSOOO1
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Malnutrition
Keywords: Cluster Randomized Trial,; Nutrition counseling,; Caretaker's knowledge; Child growth,; Prevention,; Acute malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth promotion based on child centered approach (Experimental)
  Interventions: Behavioral: Growth promotion based on child centered approach
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Growth promotion based on child centered approach — - Preventive consultations will be reorganized. From the child birth, a follow-up schedule will be establish in agreement with the mother, and the subsequent appointment will be renew at each meeting.
  Ten contacts will be organized for children under two years. During the first year, the number of contacts will be limited to 6 at birth , 2 , 3, 4 and 9 months to complete the vaccination schedule and an additional contact at 7 months to allow monitoring during the introduction of complementary foods.
  Four contacts will be held for the second year to 12, 15, 18 and 24 months to monitor the transition from complementary food to the family diet.
  - Inclusion of Child Centered growth promotion approach. During preventive consultations, specific messages according to the child age, health and nutritional status will be developed, based on scientific evidences and adapted to the experience and knowledge of health workers.
  Arms: Growth promotion based on child centered approach

SUMMARY:
Hypothesis N°1: The "children growth promotion based on approach centered on their specific needs" enhances caretakers and health workers skills, knowledge and practices on breastfeeding, complementary feeding and child care.

Hypothesis N°1: children growth promotion based on approach centered on their specific needs" approach improves children growth and health.

ELIGIBILITY:
-Inclusion Criteria: all women of childbearing age in the third trimester of pregnancy, living in the study area for at least one year at the time of the inclusion and who gave informed consent.

Exclusion Criteria:

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2341 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of acute malnutrition | 18 months

SECONDARY OUTCOMES:
Incidence of Diarrhea, fever, Acute respiratory infection | 18 months

OTHER OUTCOMES:
incidence of exclusive breastfeeding rates | 18 months
Child dietary diversity score | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé, Ouagadougou, Kadiogo, Burkina Faso